CLINICAL TRIAL: NCT05405881
Title: New Tool to Assess Proprioception of the Lower Limbs in Children With Upper Motor Neuron Lesions: Feasibility, Reliability, Validity, and Relevance for Motor Function.
Brief Title: Validity and Reliability of the PROprioception Measurement Tool (PROMT)
Acronym: PROMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Collaborators: Queen Margaret University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BASEC Nr. 2021-01373
Record Dates: First submitted 2022-05-12; First posted 2022-06-06 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Child Development; Upper Motor Neurone Lesion; Cerebral Palsy; Proprioceptive Disorders
MeSH Terms: conditions — Cerebral Palsy; Somatosensory Disorders

STUDY DESIGN:
Intervention Model Description: A cross-sectional observational psychometric study with repeated assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children with upper motor neuron lesions (Other): With the Proprioception Measurement Tool (PROMT) following modalities are assessed: joint movement sense, joint position sense, and active position sense. The child has to wear on each leg two Shimmer Sensors on the lower limb and the foot. The child sits on a table or bench, and the feet are free-hanging. A table is positioned in front of the child to place the smartphone or convertible notebook at a distance where the child can press the digital button. The table with an additional U-table platform prevents the child's view towards the legs. The duration of these three tests is 20 minutes. The comparator assessments on each level of the ICF-CY are conducted, and a feasibility questionnaire (detailed described under chapter outcome measures)
  Interventions: Other: Proprioception measurement tool
- Children without UMN lesions (developing typically) (Other): With the Proprioception Measurement Tool (PROMT) following modalities are assessed: joint movement sense, joint position sense, and active position sense. The child has to wear on each leg two Shimmer Sensors on the lower limb and the foot. The child sits on a table or bench, and the feet are free-hanging. A table is positioned in front of the child to place the smartphone or convertible notebook at a distance where the child can press the digital button. The table with an additional U-table platform prevents the child's view towards the legs. The duration of these three tests is 20 minutes. A feasibility questionnaire (detailed described under chapter outcome measures)
  Interventions: Other: Proprioception measurement tool

INTERVENTIONS:
Other: Proprioception measurement tool — No intervention, as it is a psychometric properties study

SUMMARY:
This project assesses the feasibility, reliability, and validity of the PROMT in children with a UMN lesion. The study questions are: is the newly developed PROMT a feasible, reliable, and valid tool to assess lower limb proprioception in children with UMN lesions? Does the PROMT differ between children with UMN lesion and controlled neurotypically developing peers? Further, does the proprioception modalities assessed with the PROMT correlate with motor function in this group of children?

DETAILED DESCRIPTION:
Somatosensory function is essential to all our movements and activities. This is also the case for children with Upper Motor Neuron (UMN) lesions, such as cerebral palsy or acquired brain lesions. Especially one category of somatosensory function, namely proprioception, seems to play a crucial role in motor control and motor learning. To date, no validated or reliable assessment tool exists to assess the different modalities of proprioception in children with UMN lesions. Therefore, the investigators designed an Inertial Measurement Unit's (IMU)-based outcome measure to assess three proprioception modalities. These are joint movement, joint position, and dynamic position sense. With the Unity software, the investigators have created a test setting that intuitively guides the tester and the participant through the standardised measurement procedures. The aim of this study is to investigate the feasibility, reliability, validity, and relevance in correspondence to motor function of this newly developed measurement tool.

The investigators plan to recruit 50 children with and 50 without UMN lesions. The feasibility criteria will be evaluated in the group of children with UMN lesions. The children with UMN lesions will be tested three times, twice from the same rater and once from another rater, to investigate inter-rater and test-retest reliability. To assess the relevance of this somatosensory category on motor function in children with UMN lesions, specific assessments on the body function, activity, and participation level of the international classification of functioning, disability, and health (ICF) will be performed. The aged-matched peers will be assessed once with the PROMT.

The PROMT should allow clinicians to assess lower limb proprioception in children with UMN lesions in a child-friendly manner. The analysis of the reliability results should allow to measure changes and probable association to motor function can lead us to further research questions to supplement the therapy program.

ELIGIBILITY:
Inclusion Criteria:

* neuromotor impairments due to UMN lesions (diagnoses can be, for example, cerebral palsy (CP), acquired brain injuries, myelomeningocele, hydrocephalus)
* ability to sit with or without back support for 30 minutes
* ability to stand with or without support
* ability to do some steps
* informed consent.

Exclusion Criteria:

* severe visual impairment
* surgery within the last six months with involvement of the lower limbs
* botulinum toxin injection in the lower limbs within the previous three months
* unable to communicate pain or discomfort (verbally or nonverbally)
* noncompliance
* not able to follow simple short instructions

Ages: 5 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 99 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Joint Movement Sense | Through study completion, an average of 1 year
  The child must recognise and confirm the direction of movement on the digital button, while the limb will be moved by the tester in a speed of 5-15°/second. Percentage of correct identified directions out of four trials and the angle in degree (°) until the movement detection for each trial are recorded.
Joint position sense | Through study completion, an average of 1 year
  The child has to confirm a particular position (criterion position), while the limb is moved passively. Difference of degree (°) for each criterion position (delta), and the direction of the error (overestimation or underestimation of the position) are recorded.
Active position sense | Through study completion, an average of 1 year
  The child has to confirm a particular position (criterion position), while the child moves the limb active. Difference of degree (°) for each criterion position (delta), and the direction of the error (overestimation or underestimation of the position) are recorded.

OTHER OUTCOMES:
Dynamic position sense with visual control | Through study completion, an average of 1 year
  The child has to confirm a particular position (criterion position) marked with a visual target, while the child moves the limb actively. Difference of degree (°) for each criterion position (delta), and the direction of the error (overestimation or underestimation of the position) are recorded.
Tactile localization task | Through study completion, an average of 1 year
  A tactile input with a 10-gram monofilament on the sole of the foot must be identified by the child either on a map of the foot or directly by pointing to the sole of the foot. These are scored using a 4-point scale (0 of 3 = insufficient body representation, 1 of 3 = restricted body representation, 2 of 3 = diminished body representation; 3 of 3 = good body representation). Both legs are scored separately. Output: Total score per leg.
Selective control assessment of the lower extremity (SCALE) | Through study completion, an average of 1 year
  To assess selective voluntary motor control of the lower extremity (hip, knee, upper ankle, lower ankle, and toes). Each joint is scored as 2 (normal), 1 (impaired), or 0 (unable). Both legs are scored separately. Output: Total Score (per leg).
Modified Timed Up and go Test (mTUG) | Through study completion, an average of 1 year
  The child sits on a chair and is asked to stand up, walk 3 meters and touch a target, turn around, return to the chair, and sit down. The time for the task will be recorded
Gross Motor Function Measure D&E (GMFM): | Through study completion, an average of 1 year
  The Dimension D assesses 13 tasks in a standing position, Dimension E contains 14 items of walking, running, or jumping tasks. For each Dimension, a percentage score will be evaluated.
Quality Function Measure (QFM) | 1 time-point
  To assesses the quality of gross motor function rated from a video recording of the child performing the GMFM. The QFM assesses five quality of movement attributes: alignment, co-ordination, dissociated movement, stability and weight-shift. For each GMFM-66 Stand/Walk item, the three most appropriate quality attributes have been pre-selected for scoring. Each quality attribute is scored on a 4-point response scale using item-specific response options described on the Quality FM score form
Evaluation of Disability Inventory Computer Adaptive Test (PEDI-CAT) | Through study completion, an average of 1 year
  Is a computer-adapted interview to assess daily activities, mobility, social/cognitive, and responsibility. PEDI CAT has been translated into German and shows good validity and reliability. The administration time of the short version is 10 minutes.
Functional Mobility Scale (FMS) | Through study completion, an average of 1 year
  Is a score of the gait ability in the daily environment of the children over three distances (5meter, 50meter, and 500meter). For each distance, a score between 1-6 indicates the independence of walking (higher score the more independent the child is). The sum score will be calculated. The administration of this test takes 5 minutes. It will be conducted by interviewing the parents or caregivers.
Gillette Functional Assessment Questionnaire - walking Scale (FAQ) | Through study completion, an average of 1 year
  The FAQ involves a range of walking abilities, describing various levels of mobility on a 10-level ordinal scale, with the levels differing in environment, terrains, or obstacles.
Feasibility Questionnaire | Through study completion, an average of 1 year
  Includes following items: time tracking for the preparation of the test, for each PROMT modality, the export of the data, and for evaluation. The Number of technique issues. Subject feedback of the children with UMN is assessed with a visual analogue scale (measured in millimetres; (from 0-100; where 0 means very easy/or none, and 100 means very difficult/or extreme) on perception of pain or discomfort/comfort, demand for concentration and fatigue. Rater's subjective feedback assessed with a visual analogue scale (measured in millimetres; (from 0-100; where 0 means very easy/or none, and 100 means very difficult/or extreme) on application and performance of the PROMT modalities, estimation of the comprehensibility of the test instructions for the child.

CONTACTS AND LOCATIONS:
Overall Officials: Hubertus JA van Hedel, Principal Investigator — University children's Hospital Zurich, Swiss children's Rehab
Locations (1):
- Swiss Children's Rehab, Affoltern am Albis, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marsico P, Meier L, van der Linden ML, Mercer TH, van Hedel HJA. Psychometric Properties of Lower Limb Somatosensory Function and Body Awareness Outcome Measures in Children with Upper Motor Neuron Lesions: A Systematic Review. Dev Neurorehabil. 2022 Jul;25(5):314-327. doi: 10.1080/17518423.2021.2011976. Epub 2021 Dec 6. PMID 34872425
- [Background] Prinsen CAC, Mokkink LB, Bouter LM, Alonso J, Patrick DL, de Vet HCW, Terwee CB. COSMIN guideline for systematic reviews of patient-reported outcome measures. Qual Life Res. 2018 May;27(5):1147-1157. doi: 10.1007/s11136-018-1798-3. Epub 2018 Feb 12. PMID 29435801
- [Background] Damiano DL, Wingert JR, Stanley CJ, Curatalo L. Contribution of hip joint proprioception to static and dynamic balance in cerebral palsy: a case control study. J Neuroeng Rehabil. 2013 Jun 15;10(1):57. doi: 10.1186/1743-0003-10-57. PMID 23767869
- [Background] Dijkerman HC, de Haan EH. Somatosensory processes subserving perception and action. Behav Brain Sci. 2007 Apr;30(2):189-201; discussion 201-39. doi: 10.1017/S0140525X07001392. PMID 17705910
- [Background] Palisano RJ, Hanna SE, Rosenbaum PL, Russell DJ, Walter SD, Wood EP, Raina PS, Galuppi BE. Validation of a model of gross motor function for children with cerebral palsy. Phys Ther. 2000 Oct;80(10):974-85. PMID 11002433
- [Background] Uzun Akkaya K, Elbasan B. An investigation of the effect of the lower extremity sensation on gait in children with cerebral palsy. Gait Posture. 2021 Mar;85:25-30. doi: 10.1016/j.gaitpost.2020.12.026. Epub 2020 Dec 28. PMID 33508563
- [Background] Zarkou A, Lee SCK, Prosser L, Hwang S, Franklin C, Jeka J. Foot and ankle somatosensory deficits in children with cerebral palsy: A pilot study. J Pediatr Rehabil Med. 2021;14(2):247-255. doi: 10.3233/PRM-190643. PMID 33896853
- [Background] Wingert JR, Burton H, Sinclair RJ, Brunstrom JE, Damiano DL. Joint-position sense and kinesthesia in cerebral palsy. Arch Phys Med Rehabil. 2009 Mar;90(3):447-53. doi: 10.1016/j.apmr.2008.08.217. PMID 19254610